CLINICAL TRIAL: NCT02645669
Title: Effect of a Locally Delivered Probiotic as an Adjunct To Scaling And Root Planing In The Management Of Chronic Periodontitis
Brief Title: Effect of a Locally Delivered Probiotic in Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Professor and Head, Periodontics, SVSIDS, Mahabubnagar, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/2/2014; D139406038 (Other: Dr NTR University of Health Sciences, Vijayawada, India)
Record Dates: First submitted 2015-12-21; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study site (Experimental): Scaling and Root planing (SRP) was followed by placement of S boulardii-FOS mixture
  Interventions: Procedure: Study site
- Control site (Placebo Comparator): Only Scaling and Root planing (SRP) was performed
  Interventions: Procedure: Control site

INTERVENTIONS:
Procedure: Study site — The probiotic is in the form of a lyophilized powder containing approximately 5 billion colony forming units (CFU) of the Saccharomyces boulardii. At the time of administration, the probiotic mixture was mixed with fructooligosaccharide in the ratio of 4:1 to induce growth and activity in S boulardii. This was applied after scaling and root planing.
  Arms: Study site
Procedure: Control site — Only Scaling and Root planing was done.
  Arms: Control site

SUMMARY:
Saccharomyces boulardii is commonly employed as a live non-pathogenic probiotic microbial feed or food supplement. S. boulardii reduces the secretion of key pro inflammatory cytokines and promotes the production of anti-inflammatory cytokines such as IL-10, which is pertinent in the context of pathogenic mechanisms in periodontitis.

DETAILED DESCRIPTION:
One method of altering the subgingival environment is by using probiotics. Probiotics are live microorganisms, which when administered in adequate amounts, confer a health benefit on the host by passively occupying a niche that may otherwise be colonized by pathogens. This tends to limit a pathogen's ability to bind to tissue surfaces and to produce virulence factors.8 In the past few years, probiotics have been investigated for periodontal health. Studies have shown that certain gut bacteria can exert beneficial effects in the oral cavity by inhibiting pathogenic species. Teughels et al., in a study showed that application of beneficial oral bacteria subgingivally after scaling and root planing led to a more host compatible subgingival microbiota which may also effect the promotion of a beneficial host response.10 Studies have revealed that probiotic Lactobacillus strains (L. reuteri, L salivarius, L. casei, L. acidophilus) were useful in reducing gingival inflammation and the number of black-pigmented rods, including Porphyromonas gingivalis, in the saliva and subgingival plaque. Streptococcus sanguinis & S. uberis were found to inhibit the growth of periodontopathogens & a strong negative between Aggregatibacter actinomycetemcomitans and S. sanguinis. Weissella cibaria isolates in the form of probiotic rinse possess the ability to inhibit biofilm formation, both in vitro and in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having at least one pocket ≥5 mm in each quadrant were included in the study.

Exclusion Criteria:

* Medically compromised patients and patients having received any form of surgical or non-surgical therapy in the 6 month period leading to the study were not included.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
In vitro Estimation of S. boulardii viability | up to 14 days
  S boulardii-FOS mixture was stored for 3 weeks at 25ºC for periodic analysis (upto14 days) of microorganism viability on a selective medium. Briefly, the mixture was plated on Sabouraud's agar plates at 30°C and colony forming units (CFU) were enumerated after 24 to 48 h of incubation. Colonies were expressed as total log count per mg of sample (log10 CFU/mg).
Viability of the probiotic mixture in the periodontal pocket | up to 7 days
  Viable cell count was determined by serial dilution method on Emmons' modification of Sabouraud's agar medium and colonies were expressed as total log count per ml of sample (log10 CFU/ml). Only colonies that were opaque, light brown, smooth and 2-3 mm in diameter were counted.

SECONDARY OUTCOMES:
GI | up to 6 months
  Gingivitis (Modified gingival index; MGI) was measured at baseline and up to 6 months after treatment.
PI | up to 6 months
  Plaque (Plaque index; PI) was measured at baseline and up to 6 months after treatment.
PPD | up to 6 months
  Probing pocket depth (in mm) was measured at baseline and up to 6 months after treatment.
CAL | up to 6 months
  Clinical Attachment Level (CAL) was measured at baseline and up to 6 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rampalli V Chandra, MDS;DNB, Principal Investigator — IEC, SVSIDS, Mahabubnagar
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Data will be shared after publishing the study.